CLINICAL TRIAL: NCT04883203
Title: The Effect of Vitamin D Supplementation on Recovery Delays for Non Severe COVID-19 Cases
Brief Title: The Effect of Vitamin D Supplementation on COVID-19 Recovery
Acronym: COVID-VITD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Collaborators: Loussaief Chawki (Unknown); Nissaf Ben Alaya (Unknown); Cyrine Ben Nasrallah (Unknown); Manel Ben Belgacem (Unknown); Hela Abroug (Unknown); Imen Zemni (Unknown); Manel Ben fredj (Unknown); Wafa Dhouib (Unknown)
Responsible Party: Principal Investigator, Sriha Belguith_asma, Professor preventive medicine and epidemiology, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VITD COVIDMonastir
Record Dates: First submitted 2021-04-20; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: COVID 19; Vitamin D; Recovery
MeSH Terms: conditions — COVID-19 | interventions — Solutions; Ergocalciferols; Plasmalyte A

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial with 2 parallel arms and participant masking
Who Masked: Participant
Masking Description: the intervention group will have vitamin D supplementation (200,000 IU / 1 mL of Cholecalciferol (1 ml) Oral form).
  Control group will have a placebo treatment (physiological saline).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VITD (Active Comparator): A single vial of Cholecalciferol (1 ml) (200,000 IU / 1 m), Oral form,
  Interventions: Drug: Vit-D 0.2 MG/ML Oral Solution [Calcidol]
- Placebo (Placebo Comparator): A single vial of physiological salin Oral form
  Interventions: Drug: Physiological Irrigating Solution

INTERVENTIONS:
Drug: Vit-D 0.2 MG/ML Oral Solution [Calcidol] — ARM 1 : Cholecalciferol 200,000 IU / 1 mL .
  Arms: VITD
Drug: Physiological Irrigating Solution — ARM 2 : placebo
  Arms: Placebo

SUMMARY:
The COVID-19 caused by SARS-CoV-2 has transmitted quickly as a global public health emergency. The median duration for Sars-CoV-2 carrying in COVID-19 patients was 20 days (IQR 16-28) What is the role of vitamin D supplementation on the recovery time of asymptomatic and pauci-symptomatic COVID-19 subjects? the intervention group will have vitamin D supplementation (200,000 IU / 1 ml of Cholecalciferol (1 ml) Oral form). Control group will have a placebo treatment (physiological saline).

the negative RT-PCR date will be compared in the two groups

DETAILED DESCRIPTION:
Introduction In 2020 The world is incurring coronavirus pandemic. The epidemic of the new coronavirus started in Wuhan, China, in late 2019, originally called 2019-nCoV and then COVID-19 by the World Health Organization in February 2020.

COVID-19 presented a heavy health systems burden having caused more than 170,000 deaths worldwide as of April 20, 2020. However, the treatment protocols for this infection remain controversial. It is the subject of several ongoing studies.

The use of vitamin D as a strategy to reduce the frequency and severity of respiratory infections and in particular COVID-19 must be seriously considered.

Several studies have studied the role of vitamin D in reducing the risk of viral infections. Indeed, vitamin D supplementation could be a useful measure in improving the immune response of subjects affected by the new coronavirus. This, taking into account the high prevalence of vitamin D deficiency in our country.

The beneficial effects of vitamin D on protective immunity is partly due to innate immune system action. It reduces the cytokine storm induced by the innate immune system, by decreasing the expression of pro-inflammatory cytokines and increasing that of anti-inflammatory cytokines. Vitamin D played a major role in the modulation of adaptive immunity. However, evidence on the effectiveness of vitamin D in improving the immune response of confirmed COVID-19 remains lacking.

The prolonged duration of the disease may increase the likelihood of transmission. Indeed, the R0 depends on three factors including the contact rate between individuals in the population, the probability of transmission of the infection during contact and the duration of infectiousness. The COVID-19 caused by SARS-CoV-2 has transmitted quickly as a global public health emergency. The median duration for Sars-CoV-2 carrying in COVID-19 patients was 20 days (IQR 16-28)(9).

1. Research question:

   What is the role of vitamin D supplementation on the recovery time of asymptomatic and pauci-symptomatic COVID-19 subjects?
2. Objectives of the study:

   To assess the effect of vitamin D supplementation on the duration of carriage of the COVID-19 virus in patients with SARS Cov2 with a positive control RT-PCR on day 14 of the date of confirmation of the disease.
3. Type of study:

This is a randomized clinical trial without the patient's knowledge in subjects diagnosed with COVID-19.

B. Method:

1. Study setting: this study will be carried out in the governorate of Monastir in the collective isolation center
2. Eligibility criteria: patients with SARS Cov2 and having a positive RT-PCR at control in

   * 14 days from confirmation of infection for asymptomatic subjects and
   * 7 days after the disappearance of symptoms for pauci-symptomatic subjects. Non-inclusion criteria: Pregnant women and children under the age of 18 will not be included.
3. Intervention: the intervention group will have vitamin D supplementation (200,000 IU / 1 mL of Cholecalciferol (1 ml) Oral form). Control group will have a placebo treatment (physiological saline).
4. Output: the negative RT-PCR date will be compared in the two groups.
5. Variables: we will study the socio-demographic characteristics (age, sex, level of study) and the recovery dates (dates of confirmation samples, disappearance of symptoms and control) the presence of hospitalization.
6. Sample size: for a gain of 07 days for healing, with 90% power and a 2-sided 0.05 significance level, 130 patients were required (65 in each group).

C. Allocation of interventions:

After a phone agreement, a doctor ensures the treatment distribution. D. Ethical considerations This survey will be carried out respecting the research ethical considerations: consent (free, informed, written, clear and loyal) anonymity; confidentiality; protection and assistance.

E. Study budget The Monastir University Hospital of Monastir will fund study (buying Vit D). F. Study schedule This interventional investigation will begin in July 2020. Patient monitoring will be carried out until the recovery date. (2 negative RT-PCR tests).

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID 19 and having a positive RT-PCR at control in

  * 14 days from confirmation of infection for asymptomatic subjects and
  * 7 days after the disappearance of symptoms for pauci-symptomatic subjects

Non inclusion Criteria: Pregnant women and children under the age of 18 will not be included

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D supplementation and recovery delay in COVID-19 patients | 3 months
  Delay between the first positive RT-PCR and the second negative RT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Asma Sriha Belguit, Monastir, Tunisia

REFERENCES:
- [Derived] Abroug H, Maatouk A, Bennasrallah C, Dhouib W, Ben Fredj M, Zemni I, Kacem M, Mhalla S, Nouira S, Ben Belgacem M, Nasri A, Klii R, Loussaief C, Ben Alya N, Bouanene I, Belguith Sriha A. Effect of vitamin D supplementation versus placebo on recovery delay among COVID-19 Tunisian patients: a randomized-controlled clinical trial. Trials. 2023 Feb 20;24(1):123. doi: 10.1186/s13063-023-07114-5. PMID 36803273